CLINICAL TRIAL: NCT00005225
Title: Apolipoprotein Polymorphisms and Risk of Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1104; R01HL038840 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Arteriosclerosis; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease; Coronary Disease

SUMMARY:
To determine the relative risk in a defined population of angiographically demonstrated coronary artery disease due to genetic polymorphisms at the four apolipoprotein genomic regions.

DETAILED DESCRIPTION:
BACKGROUND:

Numerous epidemiological studies have shown that the risk of coronary heart disease is strongly influenced by plasma lipid levels, especially HDL and LDL cholesterol, and their specific apolipoprotein constituents. Genetic studies have established significant heritability of these lipid components, and have also identified relatively rare major genes that result in extreme lipid values and increased risk of coronary heart disease. Geneticists have identified a number of segregating polymorphisms at the four major apolipoprotein genomic regions, using a combination of protein and DNA assays. However, in 1988 when the study was initiated, the relationship between these polymorphisms and risk of coronary heart disease had not yet been properly defined.

DESIGN NARRATIVE:

The study had a case-control design. Cases were consecutively selected from the pool of eligible Latter Day Saints Hospital patients referred for coronary angiogram. Eligibility criteria included residing in the Wasatch County or Southern Idaho counties, being healthy at the time of angiogram and having greater than 60 percent occlusion. Approximately 80-100 controls were retrospectively selected from the clinic records of the past four years. Fasting lipid profiles were defined for cases and controls in terms of total cholesterol, total triglycerides, HDL levels, LDL levels, VLDL levels, density gradient distribution of HDL-LDL subfractions, and levels of apo A-1, apo B, and apo E. The distribution of genetic polymorphisms at the four major apolipoprotein genomic regions was determined by typing all cases and controls for isoforms of apo E and apo AIV and a wide variety of DNA polymorphisms. Approximately 800 first degree relatives of cases and controls were also typed for DNA polymorphisms. Data were collected on risk factors including smoking, alcohol use, obesity, physical activity, and diet. Clinical data included medical and family history of cardiovascular disease and medication status. Multivariate statistical analysis was used to define the relative risk of coronary disease associated with segregating polymorphisms, and DNA haplotypes at these loci in conjunction with lipid profiles and risk factors. Analyses were also conducted on the extent to which the genetic segregation at these apolipoprotein genomic regions influenced the distribution of lipid profiles and whether the distribution of risk factors was influenced by the interaction of environmental risk factors such as smoking and genotypes at these regions.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-04; Study Completion 1991-03

REFERENCES:
- [Background] Marshall HW, Morrison LC, Wu LL, Anderson JL, Corneli PS, Stauffer DM, Allen A, Karagounis LA, Ward RH. Apolipoprotein polymorphisms fail to define risk of coronary artery disease. Results of a prospective, angiographically controlled study. Circulation. 1994 Feb;89(2):567-77. doi: 10.1161/01.cir.89.2.567. PMID 8313545
- [Background] Ludwig E, Corneli PS, Anderson JL, Marshall HW, Lalouel JM, Ward RH. Angiotensin-converting enzyme gene polymorphism is associated with myocardial infarction but not with development of coronary stenosis. Circulation. 1995 Apr 15;91(8):2120-4. doi: 10.1161/01.cir.91.8.2120. PMID 7697839